CLINICAL TRIAL: NCT05220267
Title: Anlotinib Plus Sintilimab as First-line Treatment for Advanced Non Clear Cell Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Director, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2021-245-02
Record Dates: First submitted 2021-12-24; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Non Clear Cell Renal Carcinoma
MeSH Terms: interventions — anlotinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib plus Sintilimab (Other): Anlotinib was taken orally (10mg mg qd, d1-14, 21 days per cycle) .Sintilimab was administered intravenously (200mg once every 3weeks).
  Interventions: Drug: Anlotinib plus Sintilimab

INTERVENTIONS:
Drug: Anlotinib plus Sintilimab — Anlotinib was taken orally (10mg mg qd, d1-14, 21 days per cycle).Sintilimab was administered intravenously (200mg once every 3weeks).

SUMMARY:
The combination of immune checkpoint inhibitors (ICIs) plus angiogenesis inhibitors has demonstrated significant anti-tumor activity in certain cancer. The goal of this study was to evaluate the efficacy and safety of sintilimab (a human programmed death-1 ICI) plus anlotinib (a multi-target tyrosine kinase inhibitor, inhibiting tumor angiogenesis and proliferative signaling) in advanced non clear cell renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily joined the study and signed informed consent;
* Aged > 18 years;
* ECOG body status score is 0 or 1,Expected survival time is greater than 3 months.
* Locally advanced or metastatic, histological confirmed, non-clear cell RCC of all subtypes. Patients must have advanced non-clear cell of one of the following subtypes: papillary, chromophobe, collecting duct carcinoma (CDC), renal medullary carcinoma (RMC), or unclassified.
* Patients must have measurable lesions as defined by the RECIST 1.1 standard;
* Adequate hematologic and end-organ function as defined by the following laboratory results obtained within 28 days prior to the first study treatment:

  1. Absolute neutrophil count (ANC) ≥1.5x 109/L
  2. Lymphocyte count ≥ 500/uL.
  3. Platelet count ≥ 80x109/L.
  4. Hemoglobin ≥ 80 g/L (patients may be transfused to meet this criterion).
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) with the following exceptions: Patients with documented liver/bone metastases should have AST and ALT ≤ 5 x ULN.
  6. Serum bilirubin ≤ 1.5 x ULN.
  7. Creatinine clearance ≥ 60 mL/min.
  8. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective forms of contraception and to continue its use 4 weeks after the last dose of anlotinib or sintilimab.
* Signed informed consent form.
* Ability and capacity to comply with study and follow-up procedures.

Exclusion Criteria:

* Those who are known to be allergic to pharmaceutical ingredients.
* Receive anti-tumor monoclonal antibody or other research drugs within 4 weeks before enrollment; have received other anti-PD-1 antibody therapy or other treatment for PD-1/PD-L1;
* Previous use of anlotinib or other angiogenesis inhibitors
* The patient has any active autoimmune disease or a history of autoimmune disease;
* There are uncontrolled heart clinical symptoms or diseases;
* Patients with congenital or acquired immune deficiency;
* Receive chemotherapy, targeted therapy, radiotherapy within 2 weeks before enrollment;
* A history of gastrointestinal perforation or major surgery within 4 weeks before enrollment;
* Overactive/venous thrombosis occurred within 6 months prior to enrollment, such as cardiovascular-cerebral vascular (including transient ischemic attack),deep vein thrombosis (except for patients who have recovered from venous catheterization due to previous chemotherapy)and pulmonary embolism;
* Those with active bleeding or bleeding tendency;
* Presence of a drug uncontrolled hypertension;
* Urine routine indicates more than urinary protein 2+;
* Correct QT interval > 470msec; if the patient has a prolonged QT interval, but the investigator's study evaluates that the prolongation is due to a cardiac pacemaker (and no other abnormalities in the heart), it is necessary to discuss with the sponsor's researcher to determine if the patient is Suitable for group study;
* Patients suspected of having other primary cancers;
* Those who are known to be allergic to pharmaceutical ingredients.
* Patients with active or chronic hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening). Patients with past/resolved HBV infection (defined as having negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. A negative HBA DNA test must be obtained in patients with positive hepatitis B core antibody prior to Cycle 1 Day 1.
* Active hepatitis C infection. Patients positive hepatitis C antibody test are eligible if PCR is negative for hepatitis C viral DNA.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | up to 2 years
  Time from treatment until disease progression or death

SECONDARY OUTCOMES:
objective response rate (ORR) | up to 2 years
  objective response rate (ORR) by RECIST1.1, the total proportion of patients with complete response (CR), partial response (PR)
disease control rate (DCR) | up to 2 years
  disease control rate (DCR)by RECIST1.1, the total proportion of patients with complete response (CR), partial response (PR) and Stable Disease(SD).
overall survival (OS) | up to 2 years
  Time from treatment until death from any cause
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] 1. Bray F,Ferlay J,Soerjomatarm I,et al.Global cancer statistics 2018:GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries[J].CA Cancer J Clin,2018,68(6):394-424. 2. Choueiri T,Motzer R.Systemic therapy for metastatic renal-cell carcinoma[J].N Engl J Med,2017,376(4):354-366 3. ESCUDIER B,EISEN T,STADLER W M,et al.Sorafenib in advanced clear cell renal-cell carcinoma[J].N Engl J Med,2007,356(2):125-134 4. MOTZER R J,HUTSON T E,TOMCZAK P,et al.Overall survival and updated results for sunitinib compared with interferon alfa in patients with metastatic renal cell carcinoma[J].J Clin Oncol,2009,27(22):3584-3590 5. Armstrong AJ, Halabi S, Eisen T, et al. Everolimus versus sunitinib for patients with metastatic non-clear cell renal cell carcinoma (ASPEN): a multicentre, open-label, randomised phase 2 trial. Lancet Oncol. 2016;17(3):378-388. 6. Nizar M Tannir, Eric Jonasch, Laurence Albiges, et al. Everolimus Versus Sunitinib Prospective Evaluation in Metastatic Non-Clear Cell Renal Cell Carcinoma (ESPN): A Randomized Multicenter Phase 2 Trial[J]. European Urology, 2016, 69(5):866-874. 7. Motzer RJ, Barrios CH, Kim TM, et al.: Phase II randomized trial comparing sequential first-line everolimus and second-line sunitinib versus first-line sunitinib and secondline everolimus in patients with metastatic renal cell carcinoma. J Clin Oncol 2014; 32:2765-2772. 8. Zhou AP,Bai Y,Song Y,et al. Anlotinib Versus Sunitinib as First-Line Treatment for Metastatic Renal Cell Carcinoma:A Randomized PhaseⅡClinical Trial[J]. Oncologist,2019,24(8):e702-e708. DOI:10.1634/theoncologist.2018-0839. 9. CHOUEIRI T K,FISHMAN M N,ESCUDIER B,et al.Immunomodulatory activity of nivolumab in metastatic renal cell carcinoma[J].Clin Cancer Res,2016,22(22):5461-5471. 10. MCDERMOTT D F,SOSMAN J A,SZNOL M,et al.Atezolizumab,an antiprogrammed death-ligand 1 antibody,in metastatic renal cell carcinoma:long-term safety,clinical activity,and immune correlates from a phase Ⅰa study[J].J Clin Oncol,2016,34(8):833-842. 11. Rini, BI; Plimack, ER; Stus, V; et al.Pembrolizumab plus Axitinib versus Sunitinib for Advanced Renal-Cell Carcinoma.[J].N Engl J Med.2019,380(12):1116-1127 12. YASUDA S,SHO M,YAMATO I,et al.Simultaneous blockade of programmed death 1 and vascular endothelial growth factor receptor 2 (VEGFR2) induces synergistic anti-tumour effect in vivo[J].Clin Exp Immunol,2013,172:500-506